CLINICAL TRIAL: NCT03033784
Title: Target Engagement for Intranasal Oxytocin in Autism Spectrum Disorders, an fMRI Dose Response Study
Brief Title: Autism Oxytocin Brain Project
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Elissar Andari, Adjunct Assistant Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00093455; P50MH100023 (NIH)
Record Dates: First submitted 2017-01-24; First posted 2017-01-27 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: Neuroscience
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Autism Spectrum Disorder (ASD) (Experimental): Male participants diagnosed with ASD will receive 12 puffs (6 in each nostril) of intranasal oxytocin (syntocinon) and placebo (assigned randomly) during 4 study visits.
  Interventions: Drug: 8 International Units (IU) of Oxytocin; Drug: 24IU of Oxytocin; Drug: 48IU of Oxytocin; Drug: Placebo
- Healthy Control (Placebo Comparator): Age matched healthy controls will receive placebo intranasal spray (12 puffs, 6 per nostril) during one study visit.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 8 International Units (IU) of Oxytocin — Participants will receive one dose of intranasal oxytocin at a dose of 8IU.
  Other Names: syntocinon
  Arms: Autism Spectrum Disorder (ASD)
Drug: 24IU of Oxytocin — Participants will receive one dose of intranasal oxytocin at a dose of 24IU.
  Other Names: syntocinon
  Arms: Autism Spectrum Disorder (ASD)
Drug: 48IU of Oxytocin — Participants will receive one dose of intranasal oxytocin at a dose of 48IU.
  Other Names: syntocinon
  Arms: Autism Spectrum Disorder (ASD)
Drug: Placebo — Participants will receive an intranasal placebo to match the oxytocin doses.

SUMMARY:
The main goal of the study is to look at the effects of intranasal oxytocin on the brain in Autism Spectrum Disorder (ASD). Oxytocin is a hormone that exists naturally in the body and the brain, affecting a wide range of social behaviors and emotions. The investigators will study the effects of different treatments (3 doses of oxytocin and one dose of placebo) on brain functional connectivity at rest in patients with ASD, using functional magnetic resonance imaging (fMRI). Investigators also seek to study how the effects of oxytocin treatment can be affected by genetic, immune and environmental factors.

DETAILED DESCRIPTION:
This study consists of investigating the effects of several doses of acute administration of intranasal oxytocin on brain activity in adults with Autism Spectrum Disorder (ASD). There is increasing evidence for the role of intranasal oxytocin (IN-OT) in enhancing social skills in ASD. Nevertheless, there is still a need of determining target engagement for oxytocin's action on brain and behavior. Here, investigators are studying the effects of different doses of IN-OT on the modulation of behavioral outcomes and neural responses in a double blind crossover study in individuals with ASD.

The aims of the research are to:

1. Study the effects of IN-OT doses on the modulation of brain functional connectivity between key socio-emotional brain regions during resting state in ASD
2. Study the effects of IN-OT doses on the blood-oxygen-level dependent (BOLD) activity of key emotional and perceptual brain networks in response to social cues (such as faces)
3. Study the effects of IN-OT on the BOLD activity of brain regions during an interactive social environment (ball game) in ASD

Investigators will compare the neuroimaging and behavioral results of individuals with ASD to control healthy males who will receive intranasal placebo. Investigators are also investigating the role of genetic factors, behavioral or clinical sub-groups of ASD, immune and environmental factors in modulating the effect of IN-OT on brain and behavior.

Participants with ASD will undergo 4 clinical visits during which they receive various randomly assigned doses of intranasal oxytocin and placebo. Both participants and the experimenter will be blind to the type of the treatment administered.

There will be only one visit for healthy controls who will all receive placebo spray. The visit for healthy controls will be conducted in a single-blind design. The experimenter will be aware that the subject is receiving placebo. However, the participant will be told that he might receive oxytocin or placebo.

ELIGIBILITY:
Inclusion Criteria for ASD Participants:

* Have an ASD diagnosis based on the Autism Diagnostic Observation Schedule (ADOS) and Autism Diagnostic Interview (ADI) criteria, gold standards of research-based autism diagnosis
* Intelligence quotient (IQ) > 70
* Normal or corrected-to-normal vision

Exclusion Criteria for ASD Participants:

* Recent occurrence of seizures (past 5 years)
* Brain damage or head trauma (can be included at discretion of PI and sponsor)
* Color blind
* Cardiovascular disease
* Presence of a severe medical problem
* Severe mental retardation
* Alcoholism or substance abuse
* Asthma (can be included at the discretion of study physician/nurse practitioner if episodes are infrequent and no active problems at time of the study)
* Migraine headaches (at the discretion of the nurse practitioner or the study physician)
* Claustrophobia (at discretion of study physician/designee/PI)
* Pacemakers, cochlear implants, surgical clips or metal fragments

Inclusion Criteria for Healthy Age-Matched Controls:

* IQ > 70
* Normal or corrected-to-normal vision

Exclusion Criteria for Healthy Age-Matched Controls:

* History of seizures
* Neurological disorder
* Current psychiatric disorder
* Previous psychiatric disorder (can be included at discretion of PI)
* Current use of psychoactive drugs
* Previous use of psychoactive drugs (can be included at discretion of PI)
* Head trauma (can be included at discretion of PI)
* Alcoholism or substance abuse
* Cardiovascular disease
* Color blind
* Asthma (can be included at the discretion of study physician/nurse practitioner if episodes are infrequent and no active problems at time of the study)
* Migraine headaches (at the discretion of the nurse practitioner or the study physician)
* Claustrophobia (at discretion of study physician/designee/PI)
* Presence of a severe medical problem
* Severe mental retardation
* Pacemakers, cochlear implants, surgical clips or metal fragments

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elissar Andari, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from a list of participants in a prior study who agreed to be contacted for future studies. Study procedures were conducted at Emory University Hospital in Atlanta, Georgia. Participant enrollment began May 10, 2017 and all study activities were completed on October 3, 2018.
Groups:
- Dose Order: Placebo, 8 International Units (IU), 24IU, 48IU: Participants with ASD randomized to receive the placebo first, followed by an 8IU of oxytocin, then 24IU dose of oxytocin, and a 48IU dose of oxytocin last.
- Dose Order: 24IU, 8IU, Placebo, 48IU: Participants with ASD randomized to receive a 24IU dose of oxytocin, followed by an 8IU of oxytocin, then the placebo, and a 48IU dose of oxytocin last.
- Dose Order: 24IU, Placebo, 8IU, 48IU: Participants with ASD randomized to receive a 24IU dose of oxytocin first, followed by the placebo, then 8IU dose of oxytocin, and a 48IU dose of oxytocin last.
- Dose Order: 48IU, Placebo, 8IU, 24IU: Participants with ASD randomized to receive a 48IU dose of oxytocin first, followed by the placebo, then an 8IU dose of oxytocin, and a 24IU dose of oxytocin last.
- Dose Order: 8IU, 24IU, Placebo, 48IU: Participants with ASD randomized to receive an 8IU dose of oxytocin first, followed by a 24IU dose of oxytocin, then the placebo, and a 48IU dose of oxytocin last.
- Dose Order: 48IU, 24IU, 8IU, Placebo: Participants with ASD randomized to receive a 48IU dose of oxytocin first, followed by a 24IU of oxytocin, then an 8IU dose of oxytocin, and the placebo last.
- Dose Order: Placebo, 48IU, 24IU, 8IU: Participants with ASD randomized to receive the placebo first, followed by a 48IU of oxytocin, then 24IU dose of oxytocin, and an 8IU dose of oxytocin last.
- Dose Order: Placebo, 24IU, 48IU, 8IU: Participants with ASD randomized to receive the placebo first, followed by a 24IU of oxytocin, then a 48IU dose of oxytocin, and an 8IU dose of oxytocin last.
- Dose Order: 48IU, 24IU, Placebo, 8IU: Participants with ASD randomized to receive a dose of 48IU of oxytocin first, followed by a 24IU of oxytocin, then the placebo, and an 8IU dose of oxytocin last.
- Dose Order: 8IU, 24IU, 48IU, Placebo: Participants with ASD randomized to receive an 8IU of oxytocin first, followed by an 24IU of oxytocin, then 48IU dose of oxytocin, the placebo last.
- Dose Order: 24IU, 48IU, 8IU, Placebo: Participants with ASD randomized to receive a 24IU dose of oxytocin first, followed by a 48IU of oxytocin, then an 8IU dose of oxytocin, and the placebo last.
- Dose Order: 48IU, 8IU, Placebo, 24IU: Participants with ASD randomized to receive a 48IU dose of oxytocin first, followed by an 8IU of oxytocin, then the placebo, and a 24IU dose of oxytocin last.
- Healthy Controls Receiving the Placebo: Healthy controls (persons without ASD) received the placebo rather than any oxytocin. The healthy controls only attended one clinical visit, per the study protocol.
Period: Overall Study
Arm/Group | Dose Order: Placebo, 8 International Units (IU), 24IU, 48IU | Dose Order: 24IU, 8IU, Placebo, 48IU | Dose Order: 24IU, Placebo, 8IU, 48IU | Dose Order: 48IU, Placebo, 8IU, 24IU | Dose Order: 8IU, 24IU, Placebo, 48IU | Dose Order: 48IU, 24IU, 8IU, Placebo | Dose Order: Placebo, 48IU, 24IU, 8IU | Dose Order: Placebo, 24IU, 48IU, 8IU | Dose Order: 48IU, 24IU, Placebo, 8IU | Dose Order: 8IU, 24IU, 48IU, Placebo | Dose Order: 24IU, 48IU, 8IU, Placebo | Dose Order: 48IU, 8IU, Placebo, 24IU | Healthy Controls Receiving the Placebo
Started (Clinical visit 1) | 9 | 2 | 4 | 4 | 3 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 19
Clinical Visit 2 | 9 | 2 | 4 | 4 | 3 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 17
Clinical Visit 3 | 9 | 1 | 4 | 4 | 3 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 0
Clinical Visit 4 | 9 | 1 | 4 | 4 | 3 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 0
Completed (Clinical Visit 4) | 9 | 1 | 4 | 4 | 3 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 17
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Anxiety related to MRI scanner | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Autism Spectrum Disorder (ASD): Male participants diagnosed with ASD received 12 puffs (6 in each nostril) of intranasal oxytocin (syntocinon) or a placebo during 4 study visits. The order in which the participant received the placebo and three different doses of oxytocin (8, 24, or 48IU) was randomly assigned.
- Healthy Control: Age matched healthy males received a placebo intranasal spray (12 puffs, 6 per nostril) during one study visit
- Total: Total of all reporting groups
Arm/Group | Autism Spectrum Disorder (ASD) | Healthy Control | Total
Number analyzed (Participants) | 32 | 19 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.97 (5.83) | 30.84 (6.50) | 29.67 (6.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 32 | 19 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 32 | 19 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 26 | 16 | 42
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 19 | 51

OUTCOME MEASURES:

1. Primary Outcome: Resting State Functional Connectivity (rsFC) Salience Network (Anterior Cingulate Cortex (ACC) and Insula Versus Visual Cortex)
Description: Investigators will study the effects of intranasal oxytocin (IN-OT) on the resting state functional connectivity between key socio-emotional and social salience brain regions using functional magnetic resonance imaging (fMRI). Resting state functional connectivity is a task-independent metric of brain activity that is based on correlations between low-frequency fluctuations of the blood oxygen level-dependent signal between several brain regions. It reflects the strength of a functional connection that is in good agreement with the underlying neuroanatomy and provides a system-level understanding of brain function. Z-scores represent the number of standard deviations from the mean of 0 and range from -3 to +3, and z-scores greater than 0 indicate greater than average resting state functional connectivity.
Time Frame: Post Intervention (Up to 40 minutes after receiving spray) at Study Visits 1, 2, 3 and 4
Population: This analysis includes participants with complete data for all visits. Two participants withdrew and data from another participant were not able to be analyzed due to technical problems during the MRI.
Measure: Mean (Standard Deviation); unit: z-scores rsFC salience-visual
Groups:
- Placebo in ASD Participants: Participants receiving the placebo
- 8IU of Oxytocin Spray: Participants receiving 8IU of oxytocin
- 24IU of Oxytocin Spray: Participants receiving 24IU of oxytocin
- 48IU of Oxytocin Spray: Participants receiving 48IU of oxytocin
- Healthy Controls Receiving Placebo: Healthy controls received the placebo spray only
Arm/Group | Placebo in ASD Participants | 8IU of Oxytocin Spray | 24IU of Oxytocin Spray | 48IU of Oxytocin Spray | Healthy Controls Receiving Placebo
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 17
z-scores rsFC salience-visual | 0.338 (0.331) | 0.400 (0.261) | 0.428 (0.248) | 0.522 (0.216) | 0.591 (0.214)

2. Primary Outcome: Blood Oxygen Level Dependent (BOLD) Activity in Response to Social Cues
Description: BOLD activity level was assessed via fMRI during completion of the face perception task (FPT) of emotional and neutral faces. BOLD scores are reported on a z-scale, with the mean, standard deviation and the minimum and the maximum. This refers to the non-thresholded z-scores that are obtained for each dose before conducting small volume correction analysis.
Time Frame: Post Intervention (Up to 70 minutes) at Study Visits 1, 2, 3, and 4
Population: This analysis includes participants with high quality images that were able to be examined. Some participants moved during the MRI resulting in distorted images.
Measure: Mean (Full Range); unit: z-scores
Arm/Group | Placebo in ASD Participants | 8IU of Oxytocin Spray | 24IU of Oxytocin Spray | 48IU of Oxytocin Spray | Healthy Controls Receiving Placebo
Number analyzed (Participants) | 26 | 28 | 29 | 25 | 17
z-scores
  Face versus Fixation, Insular Cortex | 0.347824 [-3.086408 to 2.294047] | -0.758427 [-2.614224 to 0.614738] | -0.602304 [-2.746292 to 1.613434] | 0.33747 [-2.70115 to 2.94780] | -0.540874 [-3.423316 to 2.087243]
  Face versus Fixation, Cingulate Gyrus, Anterior Division | 0.313911 [-2.50618 to 2.058421] | -0.59443 [-2.122833 to 1.013119] | -0.922999 [-2.996872 to 2.020612] | 0.03105 [-2.13638 to 2.62367] | -0.573381 [-3.103699 to 2.334144]
  Face versus Fixation, Frontal Orbital Cortex | 0.517829 [-2.3038 to 3.234023] | -0.339727 [-2.099626 to 2.850896] | 0.133334 [-2.105783 to 2.2979] | 0.51544 [-2.51943 to 3.32401] | 0.504016 [-2.080812 to 3.234903]
  Face versus Fixation, Occipital Fusiform Gyrus | 3.427291 [-0.812082 to 5.631112] | 3.556448 [-1.039342 to 6.120963] | 3.403614 [-1.445628 to 5.572412] | 3.39230 [-1.00470 to 5.80665] | 3.322934 [-0.978423 to 6.224413]
  Face versus Fixation, Left Laterobasal Amygdala | -0.003581 [-1.595989 to 2.935086] | -0.46194 [-1.821512 to 0.953573] | 0.347864 [-1.570765 to 1.521856] | 1.06647 [-1.74681 to 2.66841] | 1.341538 [-1.84355 to 3.69492]
  Face versus Fixation, Right Laterobasal Amygdala | 0.817701 [-0.488433 to 1.900966] | -0.80763 [-1.895006 to 2.793559] | 0.57701 [-0.796838 to 2.303261] | 0.989042 [-2.810703 to 3.013389] | 1.03517 [-2.307756 to 3.598735]
  Face versus Fixation, Left Accumbens | 0.324295 [-1.939803 to 1.759384] | -0.358148 [-1.451141 to 0.765259] | -0.76235 [-1.917312 to 0.928076] | -0.364131 [-1.405679 to 1.852745] | -0.859178 [-2.026179 to 1.316851]
  Face versus Fixation, Right Caudate | 0.086391 [-1.634846 to 1.335388] | -0.820473 [-2.670037 to 0.688685] | 0.536007 [-0.75045 to 2.122765] | -0.602492 [-2.543713 to 2.199534] | 0.232223 [-2.707574 to 2.410349]
  Face versus Fixation, Right Hippocampus | 0.86138 [-1.352965 to 4.348929] | -0.391579 [-1.868284 to 3.961795] | 0.194145 [-1.941021 to 4.12766] | 0.485382 [-2.754611 to 3.198802] | 0.613169 [-2.431345 to 5.088185]
  Face versus Fixation, Right Amygdala | 1.047957 [-0.621127 to 3.190074] | -0.638315 [-1.963881 to 1.061985] | 0.175908 [-1.389825 to 1.977887] | 1.302074 [-1.287299 to 2.737782] | 1.701371 [-0.697901 to 4.212626]
  Face versus Fixation, Right Accumbens | -0.316604 [-1.951857 to 0.911325] | -0.567634 [-1.789596 to 0.482181] | -0.418176 [-1.775193 to 1.027106] | -0.556553 [-1.956654 to 2.058268] | -1.532579 [-2.425838 to -0.526067]
  Face versus Fixation, Left Caudate | 0.241254 [-1.046636 to 1.514177] | -0.698518 [-1.975601 to 0.583743] | -0.041339 [-1.46476 to 1.240659] | -0.280602 [-2.330866 to 2.582442] | 0.017432 [-2.115235 to 2.203946]
  Face versus Fixation, Left Hippocampus | 0.699955 [-2.416034 to 4.59093] | -0.72534 [-1.926855 to 4.494122] | -0.033878 [-1.662279 to 4.135666] | 0.295781 [-2.781685 to 3.806] | 0.632196 [-2.667728 to 5.220928]
  Face versus Fixation, Left Amygdala | 0.221233 [-1.532993 to 1.726722] | -0.631298 [-1.901488 to 0.466238] | 0.078968 [-1.932001 to 1.317286] | 1.120718 [-1.259113 to 2.66841] | 1.65022 [-1.359844 to 3.559769]
  Happy versus Neutral, Frontal Orbital Cortex | 0.39487 [-3.876791 to 3.910739] | -0.195753 [-3.703273 to 3.396273] | 0.243287 [-2.268647 to 2.754313] | -0.625216 [-4.775246 to 3.053599] | 1.04841 [-1.382502 to 4.049732]
  Happy versus Neutral, Occipital Fusiform Gyrus | 0.684501 [-1.489766 to 2.596111] | -0.459616 [-2.702162 to 3.262832] | 0.206772 [-2.308452 to 2.749471] | 0.32432 [-3.60349 to 2.583284] | 0.795348 [-2.271818 to 3.046978]
  Happy versus Neutral, Left Accumbens | 1.430518 [-1.04353 to 2.928855] | -1.177278 [-3.294369 to 0.402549] | 0.984787 [-1.104499 to 1.914929] | -0.777588 [-3.409385 to 1.37446] | 1.059391 [-0.255741 to 2.069515]
  Happy versus Neutral, Right Caudate | 0.050791 [-1.771317 to 2.670673] | 0.132704 [-1.920536 to 2.824892] | 0.025731 [-1.896249 to 1.525611] | -0.292749 [-4.148703 to 2.352553] | 1.470176 [-0.804718 to 3.345023]
  Happy versus Neutral, Right Amygdala | 0.505732 [-1.552433 to 2.498199] | 0.040877 [-1.880963 to 2.043247] | 0.928212 [-0.763867 to 2.593808] | -0.922439 [-4.184451 to 1.664002] | 1.078819 [-0.886149 to 2.589554]
  Happy versus Neutral, Right Accumbens | 0.821772 [-0.495173 to 1.957395] | -0.129955 [-2.583269 to 2.113898] | 0.565472 [-1.049526 to 2.281018] | -0.776844 [-2.016895 to 0.594082] | 0.683166 [-0.677622 to 2.492205]
  Happy versus Neutral, Left Caudate | 0.377711 [-1.217217 to 2.477899] | 0.185452 [-1.960983 to 2.223351] | 0.58712 [-0.836157 to 2.637696] | 0.00862 [-3.291056 to 2.095994] | 1.613145 [-1.51541 to 2.993093]
  Happy versus Neutral, Left Amygdala | 0.13828 [-1.928161 to 2.436266] | -0.477983 [-3.085623 to 2.149772] | 0.561367 [-1.616188 to 2.625552] | -0.62126 [-3.873271 to 2.413952] | 1.542177 [-0.461272 to 2.734072]
  Emotion versus Neutral, Insular Cortex | 0.3329 [-2.675982 to 2.832457] | 0.462527 [-1.660037 to 2.811897] | 1.049595 [-1.273595 to 3.276281] | 0.145474 [-2.786065 to 3.332985] | 0.779819 [-2.346668 to 3.176402]
  Emotion versus Neutral, Cingulate Gyrus, Anterior Division | -0.13682 [-2.575577 to 2.913227] | 0.663003 [-1.584421 to 2.818681] | 0.89113 [-1.245631 to 3.40183] | 0.239665 [-2.31224 to 2.701743] | 1.267345 [-1.801961 to 3.327014]
  Emotion versus Neutral, Frontal Orbital Cortex | 0.444076 [-3.980701 to 4.066222] | 0.084622 [-3.465221 to 3.349507] | 0.434074 [-2.768946 to 3.143204] | -0.042926 [-3.315568 to 2.746546] | 1.116102 [-1.707134 to 3.869851]
  Emotion versus Neutral, Occipital Fusiform Gyrus | 0.547858 [-1.359913 to 3.171797] | 0.377043 [-1.896795 to 3.5329] | 0.830858 [-2.054403 to 3.167927] | 0.981023 [-1.285486 to 3.026658] | 0.967798 [-1.651371 to 3.226593]
  Emotion versus Neutral, Left Laterobasal Amygdala | -0.477913 [-2.687634 to 1.870421] | -0.085989 [-1.700797 to 2.776355] | 0.31737 [-0.895359 to 1.987475] | -0.039061 [-2.717465 to 2.075508] | 1.879398 [-1.170747 to 3.377844]
  Emotion versus Neutral, Right Laterobasal Amygdala | -0.203773 [-2.527037 to 1.933879] | -0.247527 [-2.365987 to 2.928211] | 0.482033 [-2.461489 to 2.6846] | -0.291652 [-2.0339 to 1.932592] | 1.808126 [-0.99204 to 3.175681]
  Emotion versus Neutral, Left Accumbens | 2.022323 [-0.153325 to 3.383661] | -1.05875 [-2.861125 to 0.649379] | 1.752678 [-1.440897 to 2.841185] | -0.373102 [-2.431424 to 1.562321] | 1.120372 [-0.295477 to 2.693954]
  Emotion versus Neutral, Right Caudate | -0.500704 [-2.558909 to 2.218523] | 0.916936 [-1.741694 to 3.073441] | 1.197835 [-1.169374 to 2.704396] | 0.246921 [-2.510118 to 2.197111] | 1.354862 [-0.860082 to 3.293443]
  Emotion versus Neutral, Right Hippocampus | -0.015598 [-2.428018 to 3.698757] | -0.093067 [-3.202297 to 3.501489] | 0.716515 [-2.60632 to 2.458323] | -0.011004 [-1.741691 to 1.793119] | 1.203561 [-0.834364 to 3.154893]
  Emotion versus Neutral, Right Amygdala | 0.147144 [-1.452559 to 2.200656] | 0.567225 [-0.989488 to 3.187283] | 1.009125 [-2.175977 to 2.6846] | 0.031841 [-1.604876 to 1.963714] | 1.60342 [-0.71754 to 3.148343]
  Emotion versus Neutral, Right Accumbens | 0.893013 [-0.681809 to 1.831226] | -0.307024 [-2.341113 to 2.385545] | 1.396064 [-1.57792 to 3.083594] | -0.421539 [-1.611225 to 0.916681] | 0.996732 [-0.406555 to 2.566207]
  Emotion versus Neutral, Left Caudate | -0.188575 [-2.121857 to 2.886153] | 0.971035 [-0.785839 to 2.831995] | 1.498338 [0.132905 to 3.00282] | 0.470775 [-2.18889 to 1.988801] | 1.577967 [-1.278729 to 2.883603]
  Emotion versus Neutral, Left Hippocampus | -0.057242 [-2.656764 to 2.174723] | -0.154759 [-3.093637 to 2.431969] | 0.471703 [-2.465754 to 2.760711] | 0.150852 [-2.583713 to 2.787405] | 1.211722 [-1.678622 to 3.78067]
  Emotion versus Neutral, Left Amygdala | -0.148364 [-2.244867 to 1.857259] | 0.328634 [-1.946766 to 2.938312] | 0.435674 [-1.569945 to 2.837412] | 0.659752 [-2.03181 to 2.689729] | 2.130943 [0.564661 to 3.349099]
  Negative Emotions versus Neutral, Insular Cortex | 0.078993 [-2.741794 to 2.651302] | 0.814225 [-0.964688 to 3.001415] | 1.280621 [-1.535613 to 3.649256] | 0.791272 [-1.838989 to 4.374804] | 0.869933 [-1.937001 to 2.842933]
  Negative Emotions versus Neutral, Cingulate Gyrus, Anterior Division | -0.189082 [-2.496925 to 2.594132] | 1.001123 [-0.867178 to 3.086144] | 1.064596 [-1.394323 to 3.537169] | 0.906276 [-2.548369 to 4.187496] | 1.07742 [-1.531522 to 2.899168]
  Negative Emotions versus Neutral, Occipital Fusiform Gyrus | 0.336816 [-1.818473 to 3.575764] | 0.664895 [-1.735978 to 3.302326] | 1.007465 [-2.025182 to 3.262868] | 1.263083 [-1.714918 to 3.640724] | 0.926976 [-1.643682 to 3.201217]
  Negative Emotions versus Neutral, Left Laterobasal Amygdala | -0.50816 [-2.706088 to 2.065712] | 0.11396 [-1.289767 to 3.043139] | 0.276778 [-1.192876 to 1.852493] | 0.561114 [-1.731715 to 2.259484] | 1.910744 [-0.995564 to 3.208958]
  Negative Emotions versus Neutral, Right Laterobasal Amygdala | -0.516251 [-2.699315 to 1.637606] | 0.143468 [-1.877897 to 2.858212] | 0.6247 [-2.617959 to 3.03048] | 0.230971 [-1.722826 to 2.324656] | 1.905216 [-0.464664 to 3.187876]
  Negative Emotions versus Neutral, Right Amygdala | -0.119579 [-1.766533 to 2.24458] | 0.735094 [-1.151499 to 3.192013] | 1.018509 [-2.083258 to 3.03048] | 0.554755 [-1.860525 to 2.394795] | 1.683817 [-0.853004 to 3.205723]
  Negative Emotions versus Neutral, Left Amygdala | -0.192095 [-2.406393 to 1.693166] | 0.512198 [-1.087271 to 3.282288] | 0.368682 [-1.412992 to 2.378465] | 1.091867 [-1.250699 to 2.76721] | 2.214728 [0.952909 to 3.208958]

3. Primary Outcome: Percent Change in Blood Oxygen Level Dependent (BOLD) Activity During Ball-Game Task
Description: BOLD activity in social-emotional brain regions during the perception of emotional facial videos were measured during the ball-game task. Mean percent change in contrast of parameter estimates in anatomical regions of interest are presented here. A positive value indicates increased BOLD activity while a negative value indicates decreased BOLD activity.
Time Frame: Post Intervention (up to 70 minutes) at Study Visits 1, 2, 3, and 4
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percent change in contrast
Arm/Group | Placebo in ASD Participants | 8IU of Oxytocin Spray | 24IU of Oxytocin Spray | 48IU of Oxytocin Spray | Healthy Controls Receiving Placebo
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 16
percent change in contrast
  Human Minus Computer, Negative Feedback, Left Amygdala | 0.2568 (0.0563) | 0.1379 (0.0494) | 0.1631 (0.0430) | 0.3304 (0.0658) | 0.3502 (0.0738)
  Human Minus Computer, Negative Feedback, Right Amygdala | 0.3141 (0.0621) | 0.1118 (0.0452) | 0.1979 (0.0490) | 0.3576 (0.0641) | 0.3823 (0.0796)
  Human Minus Computer, Negative Feedback, Right Laterobasal Amygdala | 0.1724 (0.0476) | 0.0921 (0.0379) | 0.0984 (0.0362) | 0.2569 (0.0666) | 0.2258 (0.0479)
  Human Minus Computer, Negative Feedback, Left Laterobasal Amygdala | 0.1512 (0.0493) | 0.0739 (0.0472) | 0.1094 (0.0417) | 0.2014 (0.0715) | 0.2717 (0.0555)
  Human Minus Computer, Negative Feedback, Ventral Anterior Insula (Sphere) | 0.1830 (0.0801) | 0.0311 (0.0574) | -0.0575 (0.0661) | 0.1866 (0.0872) | 0.0815 (0.0651)
  Human Minus Computer, Negative Feedback, Anterior Cingulate (Sphere) | 0.2604 (0.1109) | 0.0953 (0.0630) | 0.0419 (0.0497) | 0.3214 (0.0780) | 0.1406 (0.0525)
  Human Minus Computer, Positive Feedback, Anterior Cingulate (Sphere) | 0.2774 (0.0854) | 0.0996 (0.0564) | 0.1526 (0.0711) | 0.2343 (0.0696) | 0.1218 (0.0594)
  Human Minus Computer, Positive Feedback, Frontal Orbital Cortex | 0.2263 (0.0760) | 0.1338 (0.0360) | 0.1826 (0.0509) | 0.1859 (0.0575) | 0.2301 (0.0388)
  Human Minus Computer, Positive Feedback, Ventral Tegmental Area | 0.2412 (0.0738) | 0.1010 (0.0528) | 0.1889 (0.0769) | 0.1770 (0.0879) | 0.0848 (0.0607)
  Human Minus Computer, Positive Feedback, Right Caudate | 0.2540 (0.0823) | 0.1114 (0.0512) | 0.2605 (0.0753) | 0.2824 (0.0728) | 0.3004 (0.0602)
  Human Minus Computer, Positive Feedback, Right Nucleus Accumbens | 0.1139 (0.0675) | 0.1017 (0.0557) | 0.1779 (0.0575) | 0.1341 (0.0642) | 0.2092 (0.0669)
  Human Minus Computer, Positive - Negative Feedback, Anterior Cingulate (Sphere) | 0.0175 (0.0501) | 0.0084 (0.0431) | 0.1156 (0.0592) | -0.0996 (0.0443) | -0.0320 (0.0439)
  Human Minus Computer, Positive - Negative Feedback, Frontal Orbital Cortex | 0.0142 (0.0428) | 0.081 (0.0481) | 0.0826 (0.0412) | -0.0957 (0.0443) | 0.0286 (0.0359)
  Human Minus Computer, Positive - Negative Feedback, Ventral Tegmental Area | 0.1417 (0.0448) | -0.0175 (0.0391) | 0.0302 (0.0416) | -0.0940 (0.0810) | -0.0457 (0.0555)
  Human Minus Computer, Positive - Negative Feedback, Right Caudate | 0.0072 (0.0376) | 0.0205 (0.0278) | 0.1188 (0.0440) | -0.0452 (0.0527) | -0.0057 (0.0576)
  Human Minus Computer, Positive - Negative Feedback, Right Nucleus Accumbens | -0.0277 (0.0354) | 0.0528 (0.0354) | 0.1174 (0.0352) | -0.0615 (0.0417) | -0.0737 (0.0666)

4. Primary Outcome: Oxytocin Plasma Concentration
Description: Plasma concentration of oxytocin prior to administration of study intervention and after administration of study intervention will be compared between the different dose levels and placebo. Plasma concentration of oxytocin is expected to increase following administration of intranasal oxytocin.
Time Frame: Visits 1, 2, 3 and 4 (before spray and 5 minutes after spray)
Population: Only participants with ASD had blood drawn for plasma oxytocin concentrations. This analysis includes participants who provided a blood sample (one refused to give a sample).
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Placebo in ASD Participants | 8IU of Oxytocin Spray | 24IU of Oxytocin Spray | 48IU of Oxytocin Spray
Number analyzed (Participants) | 30 | 30 | 30 | 30
picogram/milliliter
  Prior to spray | 8.09 (3.97) | 11.17 (6.99) | 9.06 (3.45) | 9.72 (9.40)
  After spray | 7.75 (3.67) | 14.36 (9.28) | 17.52 (8.41) | 20.86 (12.66)

5. Secondary Outcome: Rate of Smiling During Global Clinical Interview
Description: Clinical improvements will be rated by a clinician as based on a videotaped interview conducted after the MRI scanning session. Values between the different treatment conditions will be assessed to study the effect of intranasal oxytocin on ASD at the clinical level. The improvement will be assessed based on the quality of social interaction between the experimenter and the participant, specifically as the amount of smiling behavior displayed by participants. Larger values indicate that participants are smiling more frequently.
Time Frame: Post Intervention (Up to 180 minutes after receiving spray) at Study Visits 1, 2, 3 and 4
Population: This analysis includes participants with ASD who completed the videotaped interview. One participant declined to be videotaped and is not included in this analysis.
Measure: Mean (Standard Deviation); unit: Smiles per minute
Arm/Group | Placebo in ASD Participants | 8IU of Oxytocin Spray | 24IU of Oxytocin Spray | 48IU of Oxytocin Spray
Number analyzed (Participants) | 30 | 30 | 30 | 30
Smiles per minute | 0.954 (0.724) | 0.954 (0.801) | 1.013 (0.810) | 1.015 (0.744)

6. Secondary Outcome: Milliseconds of Visual Fixation
Description: Eye gaze will be recorded via an eye tracker inside the MRI scanner during the face perception task (FPT). Visual fixation between different treatment conditions will be assessed in ASD participants.
Time Frame: Post Intervention (Up to 50 minutes) at Study Visits 1, 2, 3 and 4
Population: This analysis includes participants with ASD who had usable data for this outcome. There were difficulties with the eye tracking technology inside the MRI scanner and tracking of the pupil was not successful at all times. Healthy controls did not participate in the eye tracker portion of the study.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo in ASD Participants | 8IU of Oxytocin Spray | 24IU of Oxytocin Spray | 48IU of Oxytocin Spray
Number analyzed (Participants) | 14 | 21 | 14 | 13
milliseconds | 91786.05 (65288.71) | 82503.23 (48615.57) | 134913.00 (55067.12) | 130600.90 (66305.70)

7. Secondary Outcome: Social Learning Test (SLT) Reaction Time
Description: During the SLT, participants complete an implicit association test using faces and words. The faces that are presented in this task are partners' faces with whom participants played during the ball-game inside the MRI scanner. In this task, there are congruent blocks where neutral faces of "positive" partners are presented with friendly words and neutral faces of "negative" partners are presented with unfriendly words. During incongruent blocks, neutral faces of "positive" partners are presented with unfriendly words and neutral faces of "negative" partners are presented with friendly words. Participants match the face or the word to one of two categories. Longer reaction time indicates difficulty with selecting a category. Longer reaction time in incongruent trials signifies implicit biases were formed for the positive and negative players such that "positive" partners from the ball-game are now perceived as friendly and "negative" partners are now perceived as unfriendly.
Time Frame: Post Intervention (Up to 130 minutes) at Study Visits 1, 2, 3 and 4
Population: Among participants with autism who completed the study, two participants had outlying data and were removed from this analysis.Two healthy controls did not complete the SLT due to time constraints.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo in ASD Participants | 8IU of Oxytocin Spray | 24IU of Oxytocin Spray | 48IU of Oxytocin Spray | Healthy Controls Receiving Placebo
Number analyzed (Participants) | 29 | 29 | 29 | 29 | 15
milliseconds
  Congruent Blocks | 939.43 (605.79) | 972.08 (950.41) | 905.99 (741.22) | 896.63 (679.50) | 762.72 (335.81)
  Incongruent Blocks | 969.17 (730.30) | 960.41 (745.84) | 920.23 (622.83) | 921.90 (650.23) | 791.65 (410.01)
  Training Blocks | 790.49 (757.66) | 800.25 (922.21) | 765.53 (754.48) | 761.89 (782.89) | 655.27 (499.78)

ADVERSE EVENTS:
Time Frame: Adverse events that were potentially related to the study intervention were collected from the time of consent to participate in the study through all study visits (up to Week 5).
Description: Only treatment related adverse events were monitored. The total number of participants in each intervention is the number who were administered that treatment; one participant withdrew before being administered the 48IU dose or placebo. Healthy controls were only administered the placebo.
Groups:
- Placebo: Participants receiving the placebo
Arm/Group | Placebo | 8IU of Oxytocin Spray | 24IU of Oxytocin Spray | 48IU of Oxytocin Spray
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/32 | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/32 | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 3/48 | 4/32 | 5/32 | 5/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=48) | 8IU of Oxytocin Spray (N=32) | 24IU of Oxytocin Spray (N=32) | 48IU of Oxytocin Spray (N=31)
Lightheaded after spray (General disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Blood pressure increase (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness after spray and blood draw (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drowsiness (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Temperature increase (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Body temperature increased by 2 degrees for a few minutes
Numb left hand (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Numbing of hand while inside MRI, more than 40 minutes after spray intake
Nostril tingling after spray (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Frustration during MRI (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Frustration with game errors while in MRI, 40 minutes after the spray
Light coughing after spray (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT03033784/Prot_SAP_001.pdf
  • Informed Consent Form (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT03033784/ICF_002.pdf